CLINICAL TRIAL: NCT03313830
Title: Effect of Whey Protein Hydrolysate on Human Muscle Protein Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Meiji Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 17-0086
Record Dates: First submitted 2017-10-06; First posted 2017-10-18 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: Whey; Muscle Protein Synthesis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey Protein Hydrolysate (WPH) (Experimental): The intervention consists of Whey Protein Hydrolysate (WPH) ingestion by young healthy subjects to determine rates of muscle protein synthesis.
  Interventions: Dietary Supplement: Whey Protein Hydrolysate (WPH)
- Intact Whey Protein (WHEY) (Experimental): The intervention consists of Intact Whey Protein (WHEY) ingestion by young healthy subjects to determine rates of muscle protein synthesis.
  Interventions: Dietary Supplement: Intact Whey Protein (WHEY)

INTERVENTIONS:
Dietary Supplement: Whey Protein Hydrolysate (WPH) — Subjects will ingest WPH on one occasion.
  Arms: Whey Protein Hydrolysate (WPH)
Dietary Supplement: Intact Whey Protein (WHEY) — Subject will ingest WHEY on another occasion.
  Arms: Intact Whey Protein (WHEY)

SUMMARY:
Muscle protein synthesis can be stimulated by ingestion of protein sources, such as whey, casein or soy. Protein supplementation can be useful to restore protein turnover after exercise but also to preserve skeletal muscle mass and function in aging adults. Ingestion of large doses of essential amino acids (EAA) or certain protein supplements may be an effective strategy to induce muscle protein synthesis. However, in many cases, it may not be practical or feasible to consume a large volume of amino acids or protein required for an effective response by muscle. Several evidences show how reduced strength and muscle mass, even in early life, are predictors of early mortality which explicit the importance of developing more effective methods to improve muscle quality. Therefore, identifying the better sources of protein that have higher anabolic potency is of high significance.

The goal of this study is to determine the anabolic potency and efficacy of a new and novel Whey Protein Hydrolysate mixture (WPH) on skeletal muscle protein synthesis in healthy young subjects (age 20-35 yr). Previous studies on rats indicate WPH induces significant increases in muscle protein synthesis compared with carbohydrates or whey-amino acid mixture. WPH contains mostly peptides, which have physiological effects and could be absorbed more rapidly. Preliminary data from preclinical study has also demonstrated that WPH can stimulate muscle protein synthesis at lower doses compared with intact whey proteins. Thus, WPH could be absorbed more rapidly and may maximally stimulate muscle protein synthesis. Although there is substantial data on the individual effects of BCCA and intact protein such as whey, there have been no clinical investigations that have explored the efficacy of WPH for stimulating muscle protein synthesis in humans.

Therefore, the investigators propose that WPH will increase muscle protein synthesis.

They will compare the response of WHP to the response of WHEY when equal protein is provided in both treatments.

10 healthy subjects will be recruited and will receive both WPH and WHEY supplementation in a single blind crossover design. Muscle protein synthesis will be measured on both occasions. This acute study will allow to determine whether low dose WPH supplementation will be an effective nutritional treatment to stimulate muscle protein synthesis in young adults.

DETAILED DESCRIPTION:
The central hypothesis will be tested in 10 healthy young adults (20-35 yr). The subjects will be studied in the post-absorptive state on two different days, during which they will randomly assigned to drink a WPH or WHEY mixture.

Measures of muscle protein synthesis will be taken at baseline, one and three hours following nutrient ingestion.

The expected outcome of the proposed work is the identification of a new nutritional strategy for activating skeletal muscle protein synthesis. The findings of the proposed studies will have a positive impact, because they will allow us to translate this information into evidence-based clinical interventions to improve muscle size, strength and function and improve recovery after conditions associated with muscle wasting.

ELIGIBILITY:
Inclusion Criteria:

1. Men age 20-35 yrs
2. Stable body weight for at least 1 year
3. Able to provide written consent and understand the study requirements and procedures

Exclusion Criteria:

1. Exercise training
2. Significant heart, liver, kidney, blood, respiratory disease or thyroid issues
3. Peripheral vascular disease
4. Orthopedic injury
5. Diabetes mellitus or other untreated endocrine disease
6. Active cancer (all groups) and history of cancer
7. Acute infectious disease or history of chronic infections
8. Neurologic Injury or disease
9. Recent systemic treatment with anabolic steroids, or corticosteroids.
10. Alcohol or drug abuse
11. Tobacco use
12. Malnutrition
13. Obesity
14. Low hemoglobin levels
15. Food allergies
16. Taking dietary supplements
17. Chronic use of aspirin

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2017-10-07 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
muscle protein synthesis | change from Baseline muscle protein synthesis at 3 hours after mixture ingestion
  measure muscle protein turnover by stable isotope infusion trial

CONTACTS AND LOCATIONS:
Overall Officials: Blake Rasmussen, PhD, Principal Investigator — UTMB
Locations (1):
- UTMB, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moro T, Brightwell CR, Velarde B, Fry CS, Nakayama K, Sanbongi C, Volpi E, Rasmussen BB. Whey Protein Hydrolysate Increases Amino Acid Uptake, mTORC1 Signaling, and Protein Synthesis in Skeletal Muscle of Healthy Young Men in a Randomized Crossover Trial. J Nutr. 2019 Jul 1;149(7):1149-1158. doi: 10.1093/jn/nxz053. PMID 31095313